CLINICAL TRIAL: NCT03000725
Title: Adapting Project UPLIFT (Using Practice and Learning to Increase Favorable Thoughts) is for Hispanic Patients With Epilepsy II
Brief Title: Adapting Project UPLIFT for Hispanic Patients With Epilepsy II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-01531
Record Dates: First submitted 2016-12-20; First posted 2016-12-22 (Estimated); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UPLIFT (Active Comparator): Project UPLIFT (Using Practice and Learning to Increase Favorable Thoughts) is a home-based intervention that teaches cognitive and mindfulness skills to people with epilepsy by phone to reduce their depression and improve quality of life (QOL).
  Interventions: Behavioral: Using Practice and Learning to Increase Favorable Thoughts
- USUAL CARE (Active Comparator): Participants randomized to the UC group will receive printed educational materials on management of epilepsy in English or Spanish as preferred.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Using Practice and Learning to Increase Favorable Thoughts — Description of the UPLIFT program: Participants who choose to participate in UPLIFT will complete 8 weekly group sessions via telephone.
  Session 1: Introduction to UPLIFT/Noticing Thoughts Session 2: Checking and Changing Thoughts Session 3: Coping & Relaxing Session 4: Attention & Mindfulness Session 5: The Present as a Calm Place Session 6: Thoughts as Changeable, Thoughts as Not Fixed Session 7: Focus on Pleasure & the Importance of Reinforcement Session 8: Preventing Lapses and Giving Thanks
  Arms: UPLIFT
Behavioral: Usual Care — Participants randomized to the UC group will receive printed educational materials on management of epilepsy in English or Spanish as preferred.
  Arms: USUAL CARE

SUMMARY:
The purpose of this study is to adapt Project UPLIFT for Hispanic adults with epilepsy and depression. Project UPLIFT (Using Practice and Learning to Increase Favorable Thoughts) is a home-based intervention that teaches cognitive and mindfulness skills to people with epilepsy by phone to reduce their depression and improve quality of life (QOL); it was developed at Emory University with CDC funding. The purpose of this study is to adapt Project UPLIFT for Hispanic adults with epilepsy and depression. Project UPLIFT (Using Practice and Learning to Increase Favorable Thoughts) is a home-based intervention that teaches cognitive and mindfulness skills to people with epilepsy by phone to reduce their depression and improve quality of life (QOL); it was developed at Emory University with CDC funding.

DETAILED DESCRIPTION:
The goal of this study is to adapt Project UPLIFT for Hispanic adults with epilepsy and depression. A 2-arm randomized control trial will be conducted to evaluate the feasibility, acceptability and effects of Project UPLIFT versus usual care (UC) in Hispanic patients with epilepsy.

The specific aim of this study is: To evaluate the feasibility, acceptability and short- and long-term effects of the adapted intervention on depression and other outcomes in 72 English- and Spanish-speaking Hispanic epilepsy patients.

ELIGIBILITY:
Inclusion Criteria:

* self-identified as Hispanic
* English or Spanish speaking
* diagnosis of epilepsy for at least one year post diagnosis
* willing to participate in 8 one-hour telephone sessions every week for eight weeks.
* willing to be audio-taped
* Elevated depressive symptoms (Center for Epidemiological Studies Depression Scale (CES-D) score >13

Exclusion Criteria:

* Severe depression (CES-D > 37)
* Active suicidal ideation
* Significant cognitive impairment (evident during screening)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | 12 Months
  This measure assesses depressive symptoms in the past two weeks based on DSM-IV diagnostic criteria for major depression.

SECONDARY OUTCOMES:
Quality Of Life in Epilepsy (QOLIE-10) | 12 Months
  This measure assesses health-related quality of life for adults with epilepsy.
PROMIS-Global | 12 Months
  This 10-item measure was developed by NIH to assess physical, mental and social functioning. It is a generic rather than disease-specific measure of global health.

OTHER OUTCOMES:
Work Productivity and Activity Impairment Questionnaire (WPAI) | 12 Months
  This self-report measure assesses the impact of disease on productivity and work productivity loss due to general health or a specified health problem.
Self-Compassion Scale (SCS) | 12 Months
  This measure assesses trait levels of self-compassion, including the thoughts, emotions and behaviors associated with the various components of self-compassion.
Satisfaction with Life Scale (SWLS) | 12 Months
  This 5-item instrument measures global cognitive judgments of satisfaction with one's life.
Interpersonal Support Evaluation List (ISEL) | 12 Months
  This measure assesses the perceived availability of appraisal, belonging and tangible social support.
Five Facet Mindfulness Questionnaire Description (FFMQ) Short form | 12 Months
  This 24-item measure assesses the construct of mindfulness through five component skills: observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience.
Ruminative Responses Scale (RRS) | 12 Months
  This 22-item scale assesses cognitive responses to depressed mood.
Perceived Stress Scale (PSS-10) | 12 Months
  This 10-item measure assesses the degree to which situations in one's life are appraised as stressful or overwhelming.
Pittsburgh Sleep Quality Index (PSQI) | 12 Months
  This 19-item questionnaire assesses sleep quality over the past month.
Epilepsy Stigma Scale | 12 Months
  This 10-item measure assesses the degree to which a person believes that epilepsy is perceived as negative and interferes with relationships with others.
Healthcare Utilization | 12 Months
  This self-report questionnaire assesses the use of healthcare services (e.g., clinic visits ED visits, etc).

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Spruill, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States